CLINICAL TRIAL: NCT04950387
Title: Impact of Breathing Exercise Intervention on Breathing Sectors Engagement in Adolescent Runners During Load
Acronym: breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Bohemia (Other)
Responsible Party: Principal Investigator, Petr Bahensky, Department of Sports Studies, University of South Bohemia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LzdKtvsPfJu2014
Record Dates: First submitted 2021-06-21; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Healthy Lifestyle
Keywords: breathing pattern; breathing exercise; load; adolescents
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A randomization sequence has been generated using Randomization.org. An independent person not involved in this study made the computer-generated randomization sequence. Investigator did not know members of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants took part in breathing exercises
  Interventions: Other: Breathing exercises
- Control group (No Intervention): Participant did not take part in intervention

INTERVENTIONS:
Other: Breathing exercises — Based in yoga, common load
  Arms: Experimental group

SUMMARY:
Forty-six endurance runners, 23 males (age = 16.4±1.1) and 23 females (age=16.8±1.1) participated in our study. The contribution of abdominal, thoracic, and subclavian musculature to respiration and ventilation parameters during three different intensities on a cycle ergometer was assessed pre- and post-intervention.

DETAILED DESCRIPTION:
Subjects Forty six distance runners (14-18 years) participated in our study, 23 males (age = 16.4±1.1, height = 177.1±5.8 cm, weight = 62.4±5.8 kg) and 23 females (age = 16.8±1.1, height = 168.5±4.4 cm, weight = 55.9±4.0 kg). All participants reported a history of endur-ance running of at least six times a week for the past year. Participants were randomly al-located to an experimental group (n=23), which took part in an eight-week breathing in-tervention, or a control group (n=23), which continued training but did not carry out any breathing exercises. One participant did not complete the intervention for medical rea-sons, so was excluded from the study. The two groups, both experimental and control, followed the same training program, the only difference being that the experimental group performed breathing exercises. A randomization sequence has been generated using Randomization.org. An independent person not involved in this study made the comput-er-generated randomization sequence. The study protocol was reviewed and approved by the local Ethics Committee on October 19, 2018 (002/2018) and followed the guidelines of the World Medical Assembly Declaration of Helsinki. Written informed consent to partic-ipate was provided by guardians and verbal assessment was provided by the partici-pants.

Study design We evaluated ventilatory musculature involvement in three basic areas using a muscle dynamometer MD03 as previously described. The device is a four-channel digital muscle dynamometer that, by design, al-lows instantaneous values of muscle force to be measured in relation to time (i.e., both the force size and its dynamics can be evaluated). In general, different muscles and muscle groups on the human body can be measured. MD03 is made up of four muscle probes (we used three probes) that attach themselves to the human body with belts. The probes contain a strain transducer to a digital signal that is transmitted to a microprocessor evalua-tion unit that adjusts digital signals from the probes into a compatible form with a USB input to a notebook. Two software levels (SW1 and SW2) are part of MD03. Probe attachment sites were selected based on the kinematics of the aforementioned thoracic sectors. The first probe was placed in the lower respiratory sector on the ventral side of the level L4-5. In the middle wind sector at the level of 8.-9. ribs, on the ventral side below the sternum, a second probe was placed. A third level probe was placed in the upper respiratory sector 3.-4. ribs on the ventral side in the sternal area. Chest compression and expansion during respiration change the force applied to the individual sensors in the attached belt.

Inspiratory and expiratory forces exerted on individual probes located in the given breathing sectors were recorded for 60-sec and minute averages were determined for each probe. After 60-sec of resting data acquisition using spontaneous breathing and deep breathing, participants underwent an incremental test on a cycle ergometer (Lode, Gro-ningen, The Netherlands) and oxygen consumption, tidal volume, respiratory rate and minute ventilatory volume were continuously monitored (Metalyzer B3, Cortex, Leipzig, Germany). The testing protocol was made relative to participant body weight (i.e., W·kg-1) and began with a 4-min stage at 1 W·kg-1 followed by three, two-minute stages at progres-sive intensities (2, 3, 4 W·kg-1) and cadence was standardized to 95-100 rev·min-1. Ventilatory muscular involvement of the abdominal, thoracic, and subclavian body sectors was monitored during the last minute of each of the three submaximal intensities.

The training program lasted eight weeks. The experimental group performed breath-ing exercises daily. In the first week of the breathing intervention, training of breathing ex-ercises took place in the form of three supervised as group breathing sessions. In the following weeks, there were always two group training sessions, each last ~30 minutes. They practiced right on the schedule. On unsupervised days, participants were asked to perform exercises individually at home for at least 10 minutes. Information about the length of each individuals training session was recorded in a diary by the participant.

The set of breathing exercises was based on yoga, the aim was to activate the dia-phragm and become aware of individual breathing sectors. As such, breath training in-cluded a variety of exercises such as breathing wave training, full breathing (breathing in-to all sectors) and paced breathing (breathing in a specified rhythm). The exercises were performed in various positions, including lying down, sitting in the kneeling position, sit-ting, kneeling, and standing. All breathing was performed through the nose. At the begin-ning of the intervention, the participants breathed spontaneously, later switching to pro-longing the inspiratory and expiratory phases. They started with a 1: 1 ratio of inhale to exhale length. Gradually, the pre-exhalation and pre-exhalation phases of breath holding were included: inspiration - 6 periods, holding breath - 3 periods, exhaling - 6 periods, holding breath - 3 periods. Each of the participants adapted the exercise to their individual respiratory rate. Each of the exercises was repeated 6 times. The exercises were slow, with a deep focus on breathing, in line with the movement. Very important was the perception of the direction of movement and expansion of the chest, the behavior of the axis of the body (head, spine, pelvis), which they learned during the introductory meetings. The control group did not participate in any form of breathing training and were told to go about their lives as usual.

The follow-up testing, which was the same as the aforementioned described graded maximal test on the cycle ergometer, was performed after 8 weeks of intervention. The control group was always tested at the same time as the members of the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* healthy runners

Exclusion Criteria:

-

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change of Ratio of breathing sectors | 8 weeks
  pressure in particular sectors

SECONDARY OUTCOMES:
Change of ventilatory parameters | 8 weeks
  Tidal volume, respiratory rate, minute ventilatory volume

CONTACTS AND LOCATIONS:
Overall Officials: Petr Bahenský, Principal Investigator — University of South Bohemia in České Budějovice
Locations (1):
- University of South Bohemia, České Budějovice, Czechia

IPD SHARING:
Plan to Share IPD: No